CLINICAL TRIAL: NCT05641831
Title: A Randomized Double-Blind Placebo-Controlled Phase II Multi-Center Study of Inflammation Modification of Canakinumab to Prevent Leukemic Progression of Clonal Cytopenias of Unknown Significance (CCUS): IMPACT Study
Brief Title: Canakinumab for the Prevention of Progression to Cancer in Patients With Clonal Cytopenias of Unknown Significance, IMPACT Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uma Borate (Other)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSU-22091; NCI-2022-09409 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Clonal Cytopenia of Undetermined Significance
MeSH Terms: interventions — Specimen Handling; Biopsy; canakinumab; X-Rays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM I (canakinumab) (Experimental): Patients receive canakinumab SC on study. All patients also undergo ECHO and chest x-ray during screening, collection of blood samples during screening and follow up, and bone marrow biopsy and aspiration throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Canakinumab; Procedure: Chest Radiography; Procedure: Echocardiography; Other: Quality-of-Life Assessment
- ARM II (placebo) (Placebo Comparator): Patients receive placebo SC on study. All patients also undergo ECHO and chest x-ray during screening, collection of blood samples during screening and follow up, and bone marrow biopsy and aspiration throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Chest Radiography; Procedure: Echocardiography; Drug: Placebo Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo peripheral blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow biopsy and aspiration
Drug: Canakinumab — Given SC
  Other Names: ACZ885; Ilaris
  Arms: ARM I (canakinumab)
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Placebo Administration — Given SC
  Arms: ARM II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial tests how well canakinumab works to prevent progression to cancer in patients with clonal cytopenias of unknown significance (CCUS). CCUS is a blood condition defined by a decrease in blood cells. Blood cells are composed of either red blood cells, white blood cells, or platelets. In patients with CCUS, blood counts have been low for a long period of time. Patients with CCUS also have a mutation in one of the genes that are responsible for helping blood cells develop. The combination of genetic mutations and low blood cell counts puts patients with CCUS at a higher risk to develop blood cancers in the future. This transformation from low blood cell counts to cancer may be caused by inflammation in the body. Canakinumab is a monoclonal antibody that may block inflammation in the body by targeting a specific antibody called the anti-human interleukin-1beta (IL-1beta).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the length of time until development of a myeloid neoplasm (ie myelodysplastic syndrome [MDS], myeloproliferative neoplasm [MPN], chronic myelomonocytic leukemia [CMML], or acute myeloid leukemia [AML]) in high-risk clonal cytopenia of undetermined significance (CCUS) patients receiving canakinumab as therapeutic intervention compared to the control arm.

SECONDARY OBJECTIVES:

I. To determine the effect of canakinumab on hematological overall response rate.

II. To determine the effect of canakinumab on complete hematological response rate.

III. To determine the effect of canakinumab on response duration. IV. To determine the effect of canakinumab on overall survival. V. To determine the effect of canakinumab on mutational burden. VI. To determine the effect of canakinumab on infection-related adverse events. VII. To determine the effect of canakinumab on recovery of blood cell populations.

VIII. To determine the effect of canakinumab on cardiovascular episodes compared to a control arm.

IX. Patient reported outcomes will be collected using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C3).

EXPLORATORY OBJECTIVES:

I. To quantify changes in the bone marrow (BM) microenvironment according to immune cell constitution and cytokine levels over the course of canakinumab treatment compared to a control arm.

II. To characterize the inflammatory milieu in peripheral blood (PB) and BM samples by serial measurement and characterization of key cytokines (IL-1, IL-2, IL-6, TNF alpha and beta, and IFN-gamma), sensitivity of patient samples to these cytokines and relationships to various genes involved in clonal hematopoiesis.

III. To determine the dynamics of change in clone size of various CH genes in serial patient treatment and control samples, during the study, by a variety of assays including single cell sequencing, copy number alterations, and variant allele frequency (VAF) measurement to characterize differences in disease evolution.

IV. To collect serial measurement of immune cell populations in PB and BM of serial patient treatment and control samples, during the study, to characterize various immune cells involving both the innate and adaptive immune system including natural killer (NK) cell, T cell subsets namely effector, regulatory and memory T cells as well as various cell surface molecules such as checkpoint modulators (PD-1/PD-L1/TIM-3, LAG-3).

V. To understand the effect of global effects on the BM microenvironment of CH status/post (s/p) canakinumab treatment compared to the control patients using ribonucleic acid (RNA) sequencing and global methylation assays to further characterize unique genomic signatures in these patients.

OUTLINE: Patients are randomized to one of two arms.

ARM I: Patients receive canakinumab subcutaneously (SC) on study.

ARM II: Patients receive placebo SC on study.

All patients also undergo echocardiogram (ECHO) and chest x-ray during screening, collection of blood samples during screening and follow up, and bone marrow biopsy and aspiration throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age >= 18 with high-risk CCUS
* Must meet ALL the following criteria:

  * Unexplained, clinically meaningful cytopenias (greater than 4 months) in one or more of the following lineages: erythroid cells, neutrophils, platelets. Clinically meaningful cytopenia is institution specific and threshold may vary on age, sex, and race. Decision-making should depend upon lab values specific to the institution and supersede public works. Based upon published work, significant cytopenias are defined as the following (must meet criteria in at least one lineage):

    * Erythroid Cells:

      * Hemoglobin < 11 g/dL
    * White Blood Cells:

      * Absolute Neutrophil Count < 1800/microL and > 500/microL
    * Platelets:

      * Platelet Count < 150,000/microL and > 50,000/microL
  * MDS criteria not fulfilled
  * No other evidence of hematological malignancy
  * No or only mild (< 10%) bone marrow dysplasia
  * Blast cells < 5% detected via morphologic examination of blood and/or bone marrow smears which can also be supported by flow cytometry and/or immunohistochemical studies
  * Any of the following:

    * Isolated somatic spliceosome mutation at any VAF (SRSF2, SF3B1, U2AF1, or ZRSR2)
    * Isolated TP53 mutation greater than 5% VAF
    * At least 1 mutation in TET2, DMNT3A, or ASXL1 at any VAF coupled with at least 1 other known myeloid pathogenic somatic mutation or known pathogenic germline mutation that predisposes to myeloid malignancy as determined by next generation sequencing and bone marrow biopsy
    * A TET2, DMNT3A, or ASXL1 greater than 10% VAF coupled with another TET2, DMNT3A, or ASXL1 greater than 10% VAF
    * The presence of two or more known myeloid pathogenic somatic or germline mutations (other than TET2, ASXL1, DMNT3A, TP53, or spliceosome mutations) greater than 10% VAF
* Ability to understand and willingness to sign the written informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Patients with a history of hypertension or active hypertension are strongly encouraged to optimize blood pressure control
* Creatinine clearance greater than 45 ml/min using Cockcroft-Gault
* Total bilirubin =< 1.5 x ULN
* Aspartate transaminase (AST) < 3 x ULN
* Alanine transaminase (ALT) < 3 x ULN

Exclusion Criteria:

* Concurrent malignancy requiring active systemic therapy
* Diagnosis of MDS or any other myeloid malignancy in the patient's lifetime
* History of Hypersensitivity to canakinumab or drug of a similar class
* Active infection requiring prompt evaluation and treatment or history of recurrent infections
* Known active or recurrent hepatic disorder including cirrhosis, hepatitis B and C (via positive or indeterminate central laboratory [lab] results)
* Subjects with active tuberculosis. In subjects with a history of tuberculosis but without active tuberculosis, if the results of the evaluation require treatment per local guidelines, then the treatment should be initiated before randomization (unless otherwise required by Health Authorities or Institutional Review Board (IRB) in which case curative treatment must be completed prior to screening)
* Subjects with suspected or proven immunocompromised state or infections. If the results of this screening per local treatment guidelines or clinical practice require treatment for said infection then the patient is not eligible. Suspected or proven immunocompromised states or infections include:

  * Those with any other medical condition such as active infection, treated or untreated, which in the opinion of the investigator places the subject at an unacceptable risk for participation in immunomodulatory therapy. If in the opinion of the investigator, the patient's immunocompromised state does not pose an unacceptable risk for participation, in the absence of uncontrolled infection, and the patient does not have a history of serious infections (such as tuberculosis); then the patient may participate in this study.
  * Known history of testing positive for human immunodeficiency virus (HIV) infections. For countries where HIV status is mandatory: testing positive for HIV during screening using a local test.
  * Allogeneic bone marrow or solid organ transplant (history of any or within a certain period of time?)
  * Those requiring systemic or local treatment in doses with systemic effects e.g.:

    * Prednisone > 20 mg (or equivalent) oral or intravenous daily for > 14 days
    * Prednisone > 5 mg and =< 20 mg (or equivalent) daily for > 30 days
    * Equivalent dose of methotrexate > 15 mg weekly
    * Note: Azathioprine is allowed. Daily glucocorticoid-replacement for conditions such as adrenal or pituitary insufficiency is allowed. Topical, inhaled or local steroid use in doses that are not considered to cause systemic effects are permitted. Steroids for pre-medication related to chemotherapy as per local standard of care are permitted.
* Live or attenuated vaccination within 3 months prior to first dose of study drug (e.g. Measles/Mumps/Rubella [MMR], Yellow Fever, Rotavirus, Smallpox, etc.) and after initiation of canakinumab treatment
* Use of erythropoietin stimulating agents (ESA) or growth factors within four weeks prior to the start of the study
* Pregnant or nursing women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment and for up to 130 days after last dose of study drug. Basic contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
  * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps). For UK: with spermicidal foam/gel/film/cream/ vaginal suppository
  * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS). In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Prior to entry into this study, cisplatin-based chemotherapy, which may be toxic to the fetus, may be given. The time between the end of cisplatin-based chemotherapy and the start canakinumab/placebo treatment is variable, resulting in a variable need for continuation of highly effective contraception. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks prior to first dose of study drug. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential. If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the Informed Consent Form (ICF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to overt myeloid malignancy | From the date of randomization until the first date of overt myeloid malignancy diagnosis, assessed up to 6 years
  Will be estimated with the non-parametric Kaplan-Meier method to compute the median time as well as the percentage of study participants with a diagnosed hematologic malignancy of myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN), chronic myelomonocytic leukemia (CMML)/ acute myeloid leukemia (AML) at landmark time points (e.g., 1-year, 2-years) with corresponding 95% confidence intervals. Since this method will censor patients who die without having developed MDS/MPN/CMML/AML, we will also compute the cumulative incidence of overt myeloid malignancy that accounts for the competing risk of death in the absence of a hematologic malignancy. All randomized patients will be included in the primary endpoint analysis in the arm to which they were randomized (ie, intent-to-treat population).

SECONDARY OUTCOMES:
Hematological overall response rate | 6 month assessment
  Number of patients that achieve response divided by the number or randomized patients. Will be summarized using the method of Kaplan-Meier but also using the cumulative incidence function which would treat death in the absence of documented relapse as a completing risk.
Complete hematological response rate | 6 month assessment
  Number of patient that achieve complete response divided by the number of randomized patients. Will be summarized using the method of Kaplan-Meier but also using the cumulative incidence function which would treat death in the absence of documented relapse as a completing risk.
Duration of hematological response | From the date of first documented hematological response until the date of documented diagnosis of MDS, MPN, CMML, or AML, assessed up to 6 years
  Will be summarized using the method of Kaplan-Meier but also using the cumulative incidence function which would treat death in the absence of documented relapse as a completing risk.
Overall survival | From the date of registration until the date of death from any cause, assessed up to 6 years
  Will be estimated using the method of Kaplan-Meier and estimates at landmark time points (e.g., 1-year, 2-years) will be provided with corresponding 95% confidence intervals.
Changes in variant allele frequencies (VAFs) of somatic mutations | Up to 6 years
  Will be assessed by bone marrow biopsy (BMBx) samples with next generation sequencing (NGS). VAFs will be analyzed as a continuous variable and as the proportion of patients with at least a 50% of reduction in VAFs of somatic mutations relative to baseline using an Ion Torrent platform.
Infection-related adverse event rates | Up to 6 years
  The number of patients who have an adverse event of interest divided by the number of patients who have adverse events assessed.
Recovery of blood cell populations | Up to 6 years
  Changes in the percentages of lymphocytes and specific sub-types (ie T-cells) as well as erythroid, platelet, and neutrophil response via 2016 World Health Organization (WHO) International Working Group (IWG) hematological improvement criteria before and after therapy as assessed in bone marrow (BM) and hematological samples.
Cardiovascular episodes | Up to 6 years
  The number of patients who has a cardiovascular event of interest divided by the number of patients who have adverse events assessed.
Patient reported outcomes | Up to 6 years
  Outcomes reported using EORTC QLQ-C30 and compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Uma M Borate, MD, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (6):
- United States (6):
  - University of Miami, Miami, Florida
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu